CLINICAL TRIAL: NCT03561337
Title: Effect of Whey Protein Hydrolysate on Adaptions to Endurance Training in Well-trained Runners
Brief Title: Nutrient Supplementation Influences Mitochondria Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mette Hansen, Principal investigator, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AURunners2017
Record Dates: First submitted 2017-12-01; First posted 2018-06-19 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Performance; Nutrition; Protein

STUDY DESIGN:
Intervention Model Description: block randomized controlled intervention
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROTEIN-CARBOHYDRATE (Experimental): Intervention group receiving protein and carbohydrate supplement
  Interventions: Dietary Supplement: PROTEIN-CARBOHYDRATE
- CARBOHYDRATE (Placebo Comparator): Intervention groups receiving carbohydrate supplement
  Interventions: Dietary Supplement: CARBOHDYRATE

INTERVENTIONS:
Dietary Supplement: PROTEIN-CARBOHYDRATE — PRO before and PRO-CHO after training
  Arms: PROTEIN-CARBOHYDRATE
Dietary Supplement: CARBOHDYRATE — CHO before and after training
  Arms: CARBOHYDRATE

SUMMARY:
Twenty-four well trained runners (VO2max 60.73.7 ml O2 Kg-1 min1) completed a six week block randomized controlled intervention period. Subjects were randomly assigned to either PRO-CHO or CHO and matched in pairs for gender, age, VO2max, training and performance status. The PRO- CHO group ingested a protein beverage (0.3g kg-1) before and protein-carbohydrate beverage (0.3g protein kg-1 and 0.1g carbohydrate kg-1) after each exercise session. The CHO group ingested energy matched carbohydrate. Post-absorptive muscle biopsies were obtained pre and post intervention for analysis HAD, CS and PGC-1. Subjects completed two physical tests 6 km performance test (pre, week 1 and week 6) and aVo2max test (pre and post intervention).

ELIGIBILITY:
Inclusion Criteria:

1. maximal oxygen uptake (VO2max) of >50ml O2 kg-1 min-1 for women and >55ml O2 kg-1 min-1 for men,
2. running at least 3 times a week and
3. running being the primarily training form

Exclusion Criteria:

1. use of medicine
2. diagnosed metabolic diseases
3. injuries which hindered running and body mass index (BMI) < 25 kg m-2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | Change from week 1 to week 6
  maximal oxygen uptake (L O2/min)

SECONDARY OUTCOMES:
VDAC | Change from week 1 to week 6
  Mitochondria target measured by western blotting
CytC | Change from week 1 to week 6
  Mitochondria enzyme measured by western blotting
Performance | Change from week 1 to week 6
  6 km trial test
COX-IV | Change from week 1 to week 6
  Mitochondria target measured by western blotting
HSP60 | Change from week 1 to week 6
  Mitochondria target measured by western blotting
CD36 | Change from week 1 to week 6
  Fat transporter measured by western blotting

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University, Department for Public Health, Section for Sport Science, Aarhus
  - Sport Science, Department of Public Health, Aarhus University, Aarhus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen M, Oxfeldt M, Larsen AE, Thomsen LS, Rokkedal-Lausch T, Christensen B, Rittig N, De Paoli FV, Bangsbo J, Ortenblad N, Madsen K. Supplement with whey protein hydrolysate in contrast to carbohydrate supports mitochondrial adaptations in trained runners. J Int Soc Sports Nutr. 2020 Sep 7;17(1):46. doi: 10.1186/s12970-020-00376-3. PMID 32894140